CLINICAL TRIAL: NCT06628518
Title: FAmily Oriented Mindfulness Informed Legal Education (FAMiLE) Programme for Parent or Carers Affected by Incarceration and Improving Parenting in Nigeria: a Randomised Control Trial
Brief Title: FAmily Oriented Mindfulness Informed Legal Education (FAMiLE) Programme for Parent or Carers Affected by Incarceration and Improving Parenting in Nigeria
Acronym: FAMiLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: University of Manchester (Other); Jos University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tarela Ike, Senior Lecturer and Principal Investigator, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0003-0516-0313f
Record Dates: First submitted 2024-09-19; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Trauma; Depression; Anxiety; Parenting Intervention
Keywords: Parenting intervention; Anxiety; incarceration; family; depression; truama
MeSH Terms: conditions — Wounds and Injuries; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FAmily oriented Mindfulness informed Legal Education (FAMiLE) (Experimental): The FAmily oriented Mindfulness informed Legal Education (FAMiLE) is a four sessions intervention lasting approximately 90 minutes each. A session will be delivered weekly for 4 weeks.
  Interventions: Behavioral: FAmily oriented Mindfulness informed Legal Education (FAMiLE)
- Control - Waitlist Group (No Intervention): The control group will not receive an intervention until after the assessment periods at baseline, end of intervention and 3 months follow up before they will be administered the FAMiLE intervention.

INTERVENTIONS:
Behavioral: FAmily oriented Mindfulness informed Legal Education (FAMiLE) — The FAmily oriented Mindfulness informed Legal Education (FAMiLE) is a low-intensity intervention involving four sessions. The session will cover relevant aspects of brief mindfulness, legal education, awareness of human rights and challenges of complaint, including support. The Family oriented component will include stress management, including coping techniques and problem-solving, positive communication, behaviour modification and parenting, and a session on consolidation including sustaining gains. The intervention will also incorporate positive parenting and interactions with children.
  Arms: FAmily oriented Mindfulness informed Legal Education (FAMiLE)

SUMMARY:
Incarceration is a prevalent problem globally and in Nigeria. Its effect significantly impacts left behind parent or primary care givers and also the wellbeing of the families and children. Limited access to support has posed a constraint in effectively addressing the issues suffered by affected families in Nigeria. In addition, having a family member incarcerated could affect parenting due to factors such as anxiety, trauma, depression, poor social support, awareness of legal channels for complaint and harsh parenting to children. The implication is that it could not only have a negative impact on the affected victim but also on their parenting styles or caring responsibilities, which could be detrimental to children's development and wellbeing and resort to criminal behaviours. In essence this study seeks to examine the feasibility and acceptability of a brief FAmily oriented Mindfulness informed Legal Education (FAMiLE) intervention in comparison to the waitlist control group (who will be administered the intervention at a later date) in improving parenting, legal awareness, social cohesion, wellbeing and reducing trauma and anxiety as a result of the effect of having a family member incarcerated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Parent or carer with child(ren) or with caring responsibilities for children affected by incarceration.
* Able to provide full consent for their participation.
* A resident of the study areas (Delta, Jos or Lagos State)

Exclusion Criteria:

* Less than 18 years
* Unable to consent
* Currently undergoing severe mental health treatment
* Unable to speak the English language fluently

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-11 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
Service Satisfaction Scale | 4 weeks at the end of intervention
  A five item scale that can be used to assess and measure satisfaction, acceptability and quality of the intervention. Higher score denote positive outcomes and acceptability. Lower score denotes poor satisfaction and acceptability.

SECONDARY OUTCOMES:
Post-traumatic Stress Disorder Checklist (PCL-5) | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The PCL-5 is a 20-item self-report measure that can be used to assess the 20 DSM-5 symptoms of post traumatic stress disorder. A 5-10 point change represents reliable change (i.e., change not due to chance) and a 10-20 point change represents clinically significant change.
Generalised Anxiety Disorder (GAD-7) | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The GAD-7 is a seven item scale for screening, measuring and assessing the severity of generalised anxiety disorder. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Oslo Social Support Scale (OSSS-3) | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The scale is a 3-item self-reported measure designed for assessing and measuring the level of social support. The sum score ranges from 3 to 14, with high values representing strong levels and low values representing poor levels of social support as indicated as follows: a) 3-8 poor social support, b) 9-11 moderate social support, c) 12-14 strong social support.
Legal-informed Awareness of Complaint Channel Scale (LACCS) | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The LACCS is a 10-item scale that is designed for assessing and measuring level of awareness of complaint channels and legal rights. The scale has an overall rating of 30, with 0-7 indicating poor knowledge, 8-15 (average knowledge), 16-22 (good knowledge) and 23-30 (excellent knowledge).
Harsh Parenting Scale | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The scale is a 4 item scale use to assess harsh parenting. The scale has a rating of 20 with lower scores indicating non harsh parenting and higher scores indicating severe harsh parenting.
Parenting Stress Scale | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The PSS is an 18-item questionnaire for assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. personal development, emotional benefits,) and negative aspects of parenthood (e.g. demands on resources, and feelings of stress). Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Patient Health Questionnaire (PHQ-9) | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that will be used for screening, monitoring, measuring and assessing the severity of depression. Low scores (e.g. 0-4) indicate no depression, however, higher scores (20-27) indicates severe depression.
European Quality of Life Scale EQ-5D-5L | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The EQ-5D-5L is a 5 item scale designed to aid assessment of the generic quality of life. In the EQ-5D-5L, each dimension has five response levels: no problems (Level 1); slight (Level 2); moderate (Level 3); severe (Level 4); and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Incarceration, Stress and Parenting Scale | Baseline, 4 weeks end of intervention and 3 months post intervention.
  The scale is a 4 item scale that will be use for assessing and measuring incarceration impact, stress and parenting. The scale has an overall rating of 20 with score ranging 1-5 indicating severe stress in parenting, 5-10 indicating moderately severe stress in parenting, 11-15 mild stress in parenting and 16- 20 no stress in parenting.

IPD SHARING:
Plan to Share IPD: No
Data supporting this study cannot be made available due to the sensitive nature and ethical reasons on confidentiality.

REFERENCES:
- [Background] Ogunbosi BO, Adepoju AA, Orimadegun AE, Odaibo GN, Olaleye OD, Akinyinka OO. Challenges of caregivers and needs of children with parents in a Nigerian prison. Niger J Paediatr. 2022 Jul-Sep;49(3):240-244. PMID 36313982
- [Background] Adetunji, C.M., Gachuri, E.W. and Wanjao, J.N., (2024). Beyond Spouses' Imprisonment: Expectations of Non-incarcerated Female Partners of Inmates at Nigeria's Agodi-Ibadan Medium Correctional Facility. Journal of Sociology, Psychology and Religious, 4(1), pp.42-53.